CLINICAL TRIAL: NCT06823479
Title: Towards Organ Preservation and Cure Via Immunotherapy in Cutaneous Squamous Cell Carcinoma Patients, Normally Undergoing Morbid Curative Surgery and Radiotherapy. The MATISSE 2 Trial, an Investigator-initiated Multicentre Phase 2 Trial
Brief Title: Towards Cure Via Only Ultra-short ICB in CSCC
Acronym: MATISSE 2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UMC Utrecht (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M24MAT; 2024-516152-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-07; First posted 2025-02-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC); Cutaneous Squamous Cell Cancer; Cutaneous Squamous Cell Carcinoma of the Head and Neck; Cutaneous Squamous Cell Carcinoma
Keywords: nivolumab; opdivo; ipilimumab; yervoy; immunotherapy; intravenous; checkpoint inhibitors; neoadjuvant
MeSH Terms: interventions — Nivolumab; Immunotherapy

STUDY DESIGN:
Intervention Model Description: All patients will receive two courses of nivolumab 3 mg/kg in week 0 and week 2, and one course of ipilimumab 1 mg/kg in week 0. If a patient is a non-responder to immunotherapy, they will receive standard of care surgery (w/wo radiotherapy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant nivolumab + ipilimumab (Experimental): Intravenous neoadjuvant nivolumab 3 mg/kg in week 0 and 2 in combination with intravenous neoadjuvant ipilimumab 1 m/kg in week 0.
  Interventions: Drug: Nivolumab; Drug: Ipilumimab

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg
  Other Names: Immunotherapy
Drug: Ipilumimab — 1 mg/kg
  Other Names: Immunotherapy

SUMMARY:
The goal of this clinical trial is to determine whether cutaneous squamous cell carcinoma patients can be cured using only immunotherapy, without surgery or radiotherapy.

DETAILED DESCRIPTION:
This is an investigator-initiated phase 2 clinical trial consisting of 41 patients with stage I-IVa CSCC and an indication for morbid/extensive curative surgery. All patients will receive two courses of nivolumab 3 mg/kg in week 0 and week 2, and one course of ipilimumab 1 mg/kg in week 0. In week 5 response to immunotherapy will be evaluated using clinical examination, [18F]FDG-PET/CT imaging, regional lymph node ultrasound with FNAC (if applicable) and a multicentre multidisciplinary meeting. Non-responders will receive standard of care surgery (w/wo radiotherapy). Responders will enter a wait-and-monitor follow-up schedule in which response will be monitored every 3 months for a total of 2 years. If a patient is no longer responding to immunotherapy during follow-up they will receive standard of care surgery (w/wo radiotherapy).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* UV-related stage I to IVa CSCC with an indication for extensive or disfiguring surgery
* Stage III-IVa CSCC (T3-4N0-3M0 or T0N1-3M0) or multi-focal stage I-II CSCC
* Primary tumour site: vermillion border lip (C00.0, C00.1, C00.2), skin of lip NOS (C44.0), external ear (C44.2), skin face unspecified (ao: external lip and vestibulum nasi) (C44.3), skin scalp and neck (C44.4), overlapping lesion of skin (C44.8), primary site eyelid (C44.1), other body sites: CSCC outside head and neck area, but not vulva, anus or penis.
* World Health Organisation (WHO) performance status of 0-2
* Indication for SOC surgery with curative intent ± RT
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.5x109 /L, Platelets ≥100 x109 /L, Haemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x upper limit of normal (ULN), AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN (except patients with Gilbert Syndrome, who are eligible when total bilirubin < 3.0 mg/dL).
* Women of child-bearing potential (WOCBP) must use appropriate method(s) of contraception. They should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required time for nivolumab to undergo five x T1/2) after the last dose of the IMP.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25IU/L or equivalent units of HCG) prior to the start of ICB.
* Patients willing and able to understand the Dutch study information and protocol requirements and comply with the treatment/intervention schedule, scheduled visits, and other requirements of the study.

Exclusion Criteria:

* Distantly metastasized (stadium IVb) CSCC
* SCC localized in a mucosal surface (i.e. anus, vulva, penis or mucosal portion of lip)
* Patients for whom standard of care treatment consists of definitive (brachy)radiotherapy
* Primary or recurrent CSCC appearing in an area that has been previously irradiated
* Prior systemic therapy or immunotherapy.
* Active human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Positive test for hepatitis B virus surface antigen (HBsAg) or hepatitis C antibody (HCV Ab)
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, except: subjects with vitiligo, resolved childhood asthma/atopy, residual hypothyroidism due to an autoimmune condition requiring only hormone replacement, psoriasis not requiring systemic treatment, any condition not expected to recur in the absence of an external trigger.
* Underlying medical conditions that, in the investigator's opinion, will make the administration of the study drug hazardous or obscure the interpretation of toxicity or AEs
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids (up to 5 mg of prednisone per day is allowed)
* Patients who are pregnant or breastfeeding
* History of allergy to study drug components and/or history of severe hypersensitivity to any monoclonal antibody
* Use of other investigational drugs 30 days before study drug administration and 5 half times before study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical complete remission after only immunotherapy | From the start of immunotherapy until 24 months of follow-up
  The rate of patients with a clinical complete remission at 24 months of follow-up or at time of death prior to 24 months follow-up, whichever comes first, after only immunotherapy, without surgery, radiotherapy or maintenance immunotherapy.

SECONDARY OUTCOMES:
Rate of clinical complete remission after only immunotherapy | From the start of immunotherapy until 12 and 18 months of follow-up.
  The rate of patients with a clinical complete remission at 12 and 18 months of follow-up or at time of death prior to the specified time-point, whichever comes first, after only immunotherapy, without surgery, radiotherapy or maintenance immunotherapy
Immune-related adverse events | From the start of immunotherapy until 100 days after the last course of immunotherapy.
  The rate and type of immune-related adverse events (CTCAE v5.0, Clavien-Dindo).
Health-related quality of life (EORTC QLQ-C30) | From the start of immunotherapy until 24 months of follow-up.
  EORTC Core Quality of Life questionnaire. Rated on a Likert-type scale from one (never) to four (almost always), to evaluate different domains. Functional and global health status scales indicated towards better levels of functioning, whereas higher scores in the symptom scales demonstrated higher levels of symptoms.
Health-related quality of life (EORTC QLQ-H&N35) | From the start of immunotherapy until 24 months of follow-up.
  EORTC Head and Neck Cancer Quality of Life Questionnaire. Rated on a Likert-type scale from one (never) to four (almost always). Multi-item scales (pain, swallowing, senses, speech, social eating, social contact, and sexuality), and six symptom items (dental problems, opening mouth, dry mouth, sticky saliva, coughing, and feeling ill). Higher scores in the symptom scales demonstrated higher levels of symptoms.
Health-related quality of life (EQ5D) | From the start of immunotherapy until 24 months of follow-up.
  EuroQol Five Dimensions Health Questionnaire. Domains: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. It also includes a VAS regarding patients' "Health Today" scored between 0 and 100. Each domain will be converted into categorical values (problems vs no problems).
Health-related quality of life (CWS) | From the start of immunotherapy until 24 months of follow-up.
  Cancer worry scale. Rated on a Likert-type scale from one (never) to four (almost always), which were summed to produce a total CWS score ranging from 8 to 32, with higher scores indicating more frequent worries about cancer.
Health-related quality of life (IT) | From the start of immunotherapy until 24 months of follow-up.
  Immunotherapy questionnaire. Rated on a Likert-type scale from one (never) to four (almost always), to evaluate toxicity after immunotherapy treatment.
Health-related quality of life (sexuality questionnaire) | From the start of immunotherapy until 24 months of follow-up.
  Rated on a Likert-type scale from one (never) to four (almost always), to evaluate problems in sexual functioning.
Treatment duration | From the start of immunotherapy until the end of treatment (average 6 weeks)
  Total duration of received treatment
Treatment stops | From the start of immunotherapy until the end of treatment (average 6 weeks)
  The amount of times and the length of time the immunotherapy, surgery or adjuvant radiotherapy had to be stopped.
Disease-specific survival | From the start of immunotherapy until 2 years follow-up.
  The length of time a patient survives without death due to disease.
Recurrence-free survival | From the start of immunotherapy until 2 years follow-up.
  The length of time a patient survives without recurrent disease.
Event-free survival | From the start of immunotherapy until 2 years follow-up.
  The length of time a patient survives without recurrent disease or death of any cause.
Overall survival | From the start of immunotherapy until 2 years follow-up.
  The length of time a patient survives after treatment.
Healthcare consumption | From the start of immunotherapy until 24 months of follow-up.
  Healthcare consumption during the trial.
Cost-effectiveness | From the start of immunotherapy until 24 months of follow-up.
  The incremental cost-effectiveness ratio between quality-adjusted life years and the cost of trial-related healthcare.

OTHER OUTCOMES:
Tumor micro-environment (IHC) | From enrollment until week 5
  Temporal and spatial analyses of the TME in the lymph nodes and primary tumours will be explored using immunohistochemistry (e.g. PD-L1 expression, CPS score).
Tumor micro-environment (RNAseq) | From enrollment until week 5
  Temporal and spatial analyses of the TME in the lymph nodes and primary tumours will be explored using bulk and single-cell RNA-sequencing.
Tumor micro-environment (spatial mass cytometry) | From enrollment until week 5
  Temporal and spatial analyses of the TME in the lymph nodes and primary tumours will be explored using spatial mass cytometry.
Immune dynamics (PBMC) | From enrollment until week 5
  Temporal immune dynamics in peripheral blood will be investigated via peripheral blood mononuclear cells (PBMCs).
Immune dynamics (TCR) | From enrollment until week 5
  Temporal immune dynamics in peripheral blood will be investigated via TCR analyses of peripheral immune cells in comparison to intratumoural immune cells
ctDNA | From enrollment until week 5.
  The ctDNA in peripheral blood using CyclomicsSeq
Complement activation | From enrollment until week 5
  Complement activation, complement mediated neutrophil activation in the TME and their contribution on the immune response during neoadjuvant immunotherapy
Humoural immunity | From enrollment until week 5
  Activation of humoral immunity, and specifically treatment-induced changes in antibody production and their relation with treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Lotje Zuur, Prof. Dr., Principal Investigator — The Netherlands Cancer Institute
Locations (5):
- Netherlands (5):
  - Maastricht UMC, Maastricht, Limburg
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes